CLINICAL TRIAL: NCT06069141
Title: Comparisons of Treatment Responses of Early Syphilis to 2.4 Milliunits (MU) Single-dose Benzathine Penicillin G With or Without Doxycycline in People Living With HIV
Brief Title: Comparisons of Treatment Responses of Early Syphilis to Benzathine Penicillin G With or Without Doxycycline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital Hsin-Chu Branch (Other); Far Eastern Memorial Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Taoyuan General Hospital (Other Government); National Cheng-Kung University Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202305061MINA
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Early Syphilis, Latent, Serological Relapse After Treatment
Keywords: syphilis; rapid plasma reagin
MeSH Terms: conditions — Syphilis | interventions — Penicillin G; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single-dose BPG plus doxycycline (Active Comparator): single-dose benzathine penicillin G (2.4 MU intramuscularly once) plus doxycycline (100 mg orally twice daily for 7 days)
  Interventions: Drug: Benzathine Penicillin G; Drug: Doxycycline Capsule
- single-dose BPG (Placebo Comparator): single-dose benzathine penicillin G (2.4 MU intramuscularly once)
  Interventions: Drug: Benzathine Penicillin G

INTERVENTIONS:
Drug: Benzathine Penicillin G — Benzathine Penicillin G (2.4 MU intramuscularly once)
Drug: Doxycycline Capsule — doxycycline (100 mg orally twice daily for 7 days)
  Arms: single-dose BPG plus doxycycline

SUMMARY:
This randomized controlled superiority study will be conducted during 2023-2025. The eligible participants are adult people living with HIV (PLWH) who are newly diagnosed with early syphilis. Participants will be randomized in a 1:1 ratio to receive single-dose benzathine penicillin G (BPG) (2.4 MU intramuscularly once) plus doxycycline (100 mg orally twice daily for 7 days) or single-dose BPG. The primary outcome is serologic response, defined as a decline of rapid plasma reagin (RPR) titer by 4-fold or greater, at week 24 and week 48; and the secondary outcomes include microbiologic response of syphilis and bacterial sexually transmitted infections (STIs) assessed by nucleic-acid amplification test (NAAT) at week 4.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV (PLWH) aged ≥18 years with early syphilis
* Confirmed by a positive RPR titer with a reactive TPPA assay

Exclusion Criteria:

* PWH with RPR titers of <4
* Exposure to antibiotics with activity against T. pallidum within the preceding 4 weeks (penicillin, 3rd cephalosporin, doxycycline, macrolides)
* A known or suspected infection requiring additional treatment with an antimicrobial active against T. pallidum (penicillin, 3rd cephalosporin, doxycycline, macrolides)
* Testing positive for C. trachomatis and M. genitalium, for which doxycycline or macrolide was administered
* A history of intolerance to penicillin or doxycycline
* PLWH have already participated in this study
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Serologic response | Weeks 24 and week 48
  Either a 4-fold or greater decline in RPR titer compared to baseline or being RPR-nonreactive

SECONDARY OUTCOMES:
Microbiologic response of syphilis | Week 4
  T. pallidum PCR Ct value >38
Microbiologic response of bacterial STIs | Week 4
  negative STI PCR results
Safety of study treatment | Week 4
Adherence evaluation of tablet intake | Week 4

CONTACTS AND LOCATIONS:
Locations (9):
- Taiwan (9):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan
  - Far Eastern Memorial Hospital, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Taipei Vetetrans General Hospital, Taipei, Taiwan
  - Taoyuan General Hospital, Taoyuan District, Taiwan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chi Mei Medical Hospital, Tainan
  - National Cheng-Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No